CLINICAL TRIAL: NCT02928510
Title: Idelalisib (GS-1101)-Associated Colitis - Molecular and Cellular Mechanisms Research Proposal
Brief Title: Mechanisms of Idelalisib-Associated Diarrhea in Patients With Relapsed Chronic Lymphocytic Leukemia, Indolent Non-hodgkin Lymphoma, or Small Lymphocytic Lymphoma
Status: Terminated | Type: Observational
Why Stopped: withdrawn by sponsor
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 15-001217; NCI-2016-01002 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-001217 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2016-08-12; First posted 2016-10-10 (Estimated); Last update posted 2021-07-14 (Actual); Status verified 2021-05

CONDITIONS: Absence of Signs or Symptoms; B-Cell Non-Hodgkin Lymphoma; Digestive System Signs and Symptoms; Indolent Adult Non-Hodgkin Lymphoma; Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Chronic Lymphocytic Leukemia; Recurrent Indolent Adult Non-Hodgkin Lymphoma; Recurrent Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Signs and Symptoms, Digestive; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Colonoscopy; idelalisib; Restraint, Physical; Sigmoidoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool and biopsies from sigmoidoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Basic Science (biospecimen collection, idelalisib): Patients receive a physical examination during visit 1. A stool sample, blood sample, and 6 biopsies are collected at visit 2, and patients undergo a flexible fiberoptic sigmoidoscopy. Patients receive idelalisib PO twice daily BID after visit 2. Treatment continues in the absence of disease progression or unacceptable toxicity. A third research visit occurs upon development of idelalisib-associated diarrhea/colitis symptoms. Patients with diarrhea/colitis symptoms undergo a full colonoscopy and collection of stool and blood samples. Control patients with no diarrhea/colitis symptoms undergo all needed tests and assessments including a flexible fiberoptic sigmoidoscopy and collection of stool and blood samples. All patients undergo optional biospecimen collection at the time of disease progression.
  Interventions: Procedure: Biospecimen Collection; Procedure: Colonoscopy; Procedure: Colposcopic Biopsy; Drug: Idelalisib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Procedure: Physical Examination; Procedure: Sigmoidoscopy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo biospecimen collection
Procedure: Colonoscopy — Undergo colonoscopy
Procedure: Colposcopic Biopsy — Undergo colposcopic biopsy
Drug: Idelalisib — Given PO
  Other Names: CAL-101; GS-1101; Phosphoinositide-3 Kinase Delta Inhibitor CAL-101; Zydelig
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Procedure: Physical Examination — Undergo physical examination
  Other Names: Assessment; Physical; Physical Assessment; PHYSICAL EXAM
Procedure: Sigmoidoscopy — Undergo sigmoidoscopy
  Other Names: Proctosigmoidoscopy

SUMMARY:
This research trial studies the mechanisms of idelalisib-associated diarrhea in patients with chronic lymphocytic leukemia, indolent non-hodgkin lymphoma, or small lymphocytic lymphoma that has come back after a period of improvement. The cancer treatment drug idelalisib triggers diarrhea in some patients. Studying stool, blood, and tissue samples in the lab from patients who are given idelalisib may help doctors learn more about the side effects and may help to treat them in future patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore the cellular and molecular mechanisms of idelalisib-induced diarrhea/colitis in relapsed chronic lymphocytic leukemia (CLL), relapsed indolent non-hodgkin lymphomas (iNHL), or relapsed small lymphocytic lymphoma (SLL).

II. To further understand the mechanism of action (MOA) of idelalisib in context of the nodal microenvironment and the possible involvement of the immune system in idelalisib's anti-lymphoma activity.

OUTLINE:

Patients receive a physical examination during visit 1. A stool sample, blood sample, and 6 biopsies are collected at visit 2, and patients undergo a flexible fiberoptic sigmoidoscopy. Patients receive idelalisib orally (PO) twice daily (BID) after visit 2. Treatment continues in the absence of disease progression or unacceptable toxicity. A third research visit occurs upon development of idelalisib-associated diarrhea/colitis symptoms. Patients with diarrhea/colitis symptoms undergo a full colonoscopy and collection of stool and blood samples. Control patients with no diarrhea/colitis symptoms undergo all needed tests and assessments including a flexible fiberoptic sigmoidoscopy and collection of stool and blood samples. All patients undergo optional biospecimen collection at the time of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Food and Drug Administration (FDA)-approved indications for idelalisib of relapsed, histologically confirmed B-cell indolent non-hodgkin lymphoma (iNHL) or chronic lymphocytic leukemia (CLL)
* For iNHL: measureable nodal disease, defined as the presence of >= 1 nodal lesion that measures >= 2 cm in a single dimension as assessed by computed tomography (CT) or magnetic resonance imaging (MRI)
* Discontinuation of all other therapies (including radiotherapy or chemotherapy) for the treatment of iNHL >= 3 weeks before initiation of study treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Absolute neutrophil count > 750
* Platelets > 50,000
* Total bilirubin < 2 X institutional upper limit of normal (ULN)
* Aspartate transaminase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/ alanine transferase (ALT) serum glutamate pyruvate transaminase (SPGT) < 3 X institutional ULN
* Creatinine < 2 X institutional ULN
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent; all patients must have signed, witnessed informed consent prior to registration

Exclusion Criteria:

* Prior exposure to idelalisib
* Known histological transformation from iNHL to diffuse large B-cell lymphoma or Richter's Transformation for CLL
* Ongoing treatment with any other investigational agents
* Known central nervous system (CNS) involvement of lymphoma (CNS staging not required)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to idelalisib
* Uncontrolled inter-current illnesses including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known human immunodeficiency virus (HIV) infection (HIV testing not required)
* Known John Cunningham (JC) virus infection and/or progressive multifocal leukoencephalopathy (PML)
* Clinically active hepatitis A, B, or C infections
* NOTE: Patients with chronic hepatitis C virus (HCV) or hepatitis B virus (HBV) infection may enroll if other laboratory criteria are met; those with HBV surface antigen positivity may enroll only if maintained on appropriate suppressive antiviral therapy for the duration of enrollment in the trial
* Pregnancy or active nursing of an infant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from relapsed chronic lymphocytic leukemia (CLL), relapsed indolent Non-Hodgkin lymphomas (iNHL), or relapsed small lymphocytic lymphoma (SLL) will be enrolled in the UCLA Lymphoma Program and they will be receiving Idelalisib/Zydelig as the standard care treatment are potentially eligible for this specimen collection study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Cellular mechanisms of idelalisib-induced diarrhea/colitis assessed by a number of tests in order to provide variability in comparisons for the units of measure. | Up to 11 years
The Mechanism of Action (MOA) of idelalisib will be assessed with a number of tests in order to provide variability in comparisons for the units of measure. | Up to 11 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hommes, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States